CLINICAL TRIAL: NCT00791856
Title: An Open-label, Multiple-dose, Randomized, Two-period Crossover Study to Assess Bioequivalence of the 300 Mcg/Day Testosterone Reduced-size Patch (14 cm2) Relative to the 300 Mcg/Day Testosterone Reference Patch (28 cm2)
Brief Title: Bioequivalence of Testosterone Reduced-size Patch Relative to the Testosterone Reference Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2007016
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 28 cm2 testosterone patch
  Interventions: Drug: testosterone
- 2 (Experimental): 14 cm2 testosterone patch
  Interventions: Drug: testosterone

INTERVENTIONS:
Drug: testosterone — 28 cm2 testosterone patch, each patch is on for 4 days, 3 patches are used
  Arms: 1
Drug: testosterone — 14 cm2 testosterone patch, each patch is on for 4 days, 3 patches are used
  Arms: 2

SUMMARY:
This is an open-label, multiple-dose, randomized, two-period crossover bioequivalence study in approximately 110 surgically or naturally postmenopausal women on stable hormone therapy (i.e., estrogen for surgically postmenopausal women or a continuous regimen of estrogen plus progestin for naturally postmenopausal women) restricted to approved oral or transdermal regimens only, or not on concomitant hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* be a surgically postmenopausal female between 20 and 70 years of age who had a hysterectomy and bilateral oophorectomy at least 6 months prior to screening, or be a healthy naturally postmenopausal female between 50 and 70 years of age who had experienced amenorrhea for at least 12 months prior to screening;
* be in good general health based on medical history, physical examination, and laboratory evaluation;
* have had a mammogram, with no clinically significant abnormalities, within the preceding 12 months in subjects > 40 years of age;
* be on a stable dose of approved hormone therapy restricted to oral or transdermal regimens (vaginal products are not acceptable) for a period of at least 12 weeks prior to screening:

  * estrogen only for surgically postmenopausal women, or
  * estrogen only for naturally postmenopausal women who have been hysterectomized, or
  * a continuous regimen of estrogen plus progestin for naturally postmenopausal women who have not been hysterectomized

or not be on any hormone therapy (having stopped hormone therapy at least 12 weeks prior to screening;

Exclusion Criteria:

* have any uncontrolled acute diseases or had a major surgical operation requiring hospitalization within 1 month of screening;
* have uncontrolled or chronic diseases, such as hypertension (with diastolic blood pressure > 95 mm Hg on medication), systemic lupus erythematosus, or rheumatoid arthritis;
* have a history of myocardial infarction, bypass surgery, stroke, pulmonary embolism, or deep vein thrombosis;
* have a history of cancer within the last 5 years (except for basal cell carcinoma with a documented 6 month remission), abnormal vaginal bleeding, or tuberculosis;
* have uncontrolled diabetes mellitus with HbA1C > 7.5% (Note: only subjects who have diabetes mellitus or a fasting serum glucose level at the screening visit above the laboratory's upper limit of normal for the reference range will have HbA1C tested prior to randomization.);
* have any abnormal clinical laboratory values at screening assessed as clinically significant by the Investigator;
* have a serum thyroid stimulating hormone (TSH) value outside the normal laboratory range, confirmed by free T4 levels outside the normal laboratory range;
* have current severe dermatological problems (e.g., severe or cystic acne), including concomitant skin disease or a history of drug-induced contact dermatitis;
* have participated in a cumulative irritation test within the past 12 weeks, or have a known or suspected hypersensitivity or allergy to any transdermal systems including components of the patches used in this study;
* currently use or have a history of any androgen treatment within 6 months prior to screening, or use dehydroepiandrosterone 25 mg per day, or St. John's Wort within 4 weeks prior to baseline. Due to the large number of herbal remedies available, all other herbal supplements will be reviewed by the Sponsor during screening;

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of two testosterone patches based on baseline-corrected (AUCτ) and baseline-corrected maximum serum concentrations of total testosterone and free testosterone at steady-state | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Angela X Qu, MD, MS, Study Director — Procter and Gamble
Locations (4):
- United States (4):
  - Antonio Pizarro, MD, Fort Myers, Florida
  - Maria J Gulierrez, MD, Miramar, Florida
  - David R Mathews, MD, Overland Park, Kansas
  - Robert J Schwab, MD, Omaha, Nebraska